CLINICAL TRIAL: NCT05864118
Title: A Comparative Evaluation of Specimen Adequacy of a Traditional Nasopharyngeal Swab as Compared to Nasopharyngeal Saline Wash, Saliva, and Serum to Test for Respiratory Viruses and Antibody Response
Brief Title: Comparison of Nasopharyngeal Swab v. Nasopharyngeal Saline Wash or Saliva Collection in Testing for Respiratory Viruses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0777-22-EP
Record Dates: First submitted 2023-04-28; First posted 2023-05-18 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Tract Infections
Keywords: Adenovirus; Coronavirus 229E; Coronavirus HKU1; Coronavirus NL63; Coronavirus OC43; Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2); Human Metapneumovirus; Human Rhinovirus/Enterovirus; Influenza A virus; Influenza A virus A/H1; Influenza A virus A/H3; Influenza A virus A/H1-2009; Influenza B virus; Parainfluenza virus 1; Parainfluenza virus 2; Parainfluenza virus 3; Parainfluenza virus 4; Respiratory syncytial virus; Bordetella parapertussis; Bordetella pertussis; Chlamydia pneumoniae; Mycoplasma pneumoniae
MeSH Terms: conditions — Respiratory Tract Infections; Adenoviridae Infections; Enterovirus Infections | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Intervention Model Description: Adult emergency department patients receiving nasopharyngeal swab for respiratory viral testing meet inclusion criteria and will be asked to provide up to 4 study specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Saliva passive drool (Experimental): Participant is asked to spit saliva, through a straw, into a micro centrifuge tube. This specimen will undergo respiratory pathogen panel PCR testing and COVID-19 antibody testing.
  Interventions: Diagnostic Test: Respiratory pathogen panel PCR test; Diagnostic Test: COVID-19 antibody test
- Oral Capsule saliva (Experimental): Participant is asked to chew on a study device (Oral Capsule) with their molar teeth which will draw saliva into the device's internal specimen chamber. This specimen will undergo respiratory pathogen panel PCR testing and COVID-19 antibody testing.
  Interventions: Diagnostic Test: Respiratory pathogen panel PCR test; Diagnostic Test: COVID-19 antibody test
- NP saline wash by study device (Experimental): Participant will receive a nasopharyngeal wash with sterile saline. The irrigation saline is recollected into the device's internal specimen chamber. This specimen will undergo respiratory pathogen panel PCR testing and COVID-19 antibody testing.
  Interventions: Diagnostic Test: Respiratory pathogen panel PCR test; Diagnostic Test: COVID-19 antibody test
- Blood by standard finger stick method (Experimental): Participant is asked to provide approximately 60 uL of blood via a capillary finger stick. This specimen will undergo COVID-19 antibody testing.
  Interventions: Diagnostic Test: COVID-19 antibody test

INTERVENTIONS:
Diagnostic Test: Respiratory pathogen panel PCR test — Respiratory pathogen panel PCR test and COVID-19 antibody test.
  Arms: NP saline wash by study device; Oral Capsule saliva; Saliva passive drool
Diagnostic Test: COVID-19 antibody test — COVID-19 antibody test

SUMMARY:
Respiratory tract infections (RTIs) are prevalence community diseases and is the third leading cause of death worldwide. Rapid diagnosis of RTIs is essential as it drives decision points such as treatment, disposition, and containment. According to recent CDC (The Centers for Disease Control and Prevention) updates, nasopharyngeal swabbing is the preferred method of specimen collection for most RTIs such as SARS-COV-2. This process is invasive and traumatizing for patients as it requires probing (20 seconds) of the posterior nasopharynx with swab applicator. In some cases, this procedure has resulted in pain and injury. Because of the invasive nature of the procedure, patients often refuse testing or withdraw during the collection process resulting in inadequate specimen procurement. The study principle investigators (PI) have developed 2 novel specimen collection devices: 1) nasopharyngeal wash collection device (NP wash device) and 2) saliva collection device (the Oral Capsule). Both devices are designed for ease of use either by a healthcare professional or a patient. The benefits of such collection devices include 1) minimizing the invasive nature of the procedure because a swab applicator is not utilized and 2) minimizing infection risk to healthcare professional because the study devices can be self-administered when applicable. The study will enroll 1000 participants from a pool of patients presenting to the Nebraska Medicine Emergency Department (ED) who received a nasopharyngeal (NP) swab viral PCR test as part of their ED work up. Enrolled patients will be asked to provide four total specimens: 1) a saliva drool specimen, 2) a saliva Oral Capsule specimen, 3) a NP wash specimen, and 4) a finger stick serum specimen. Patients are able to opt out of any specimen collection method. Study specimens 1, 2, 3 will undergo a respiratory pathogen panel (RPP) PCR test and COVID-19 antibody testing. Study specimen 4 will undergo COVID-19 antibody testing and will function as a serum control for antibody detection.

DETAILED DESCRIPTION:
Respiratory tract infections (RTIs) are high prevalence community diseases and is the third leading cause of death worldwide. It is estimated that a new infectious disease emerges at a rate of one per year, making early disease detection critically important. Within the past few decades, we have seen an increase in cases of novel respiratory illnesses such as SARS (severe acute respiratory syndrome), H1N1 (Swine Influenza), MERS (Middle East respiratory syndrome), and SARS-COV-2 (severe acute respiratory syndrome coronavirus 2). Rapid diagnosis of RTIs is essential to the management of patients experiencing respiratory symptoms as it drives decision points such as treatment and disposition. There are currently millions of confirmed SARS-COV-2 cases globally. This number is likely underreported given the limitations and barriers to confirmatory testing. This problem is compounded by other RTIs such as influenza and rhinovirus, which are also tested via a nasopharyngeal swab specimen. According to recent updates from the CDC, nasopharyngeal swabbing is the preferred method of specimen collection for SARS-COV-2. The nasopharyngeal swab method is also commonly used in the testing of other viral pathogens such as influenza, respiratory syncytial virus (RSV), rhinovirus, and human parainfluenza. This process can be somewhat invasive and traumatizing for patients as it requires probing (10-20 seconds) of the posterior nasopharynx with a stiff swab applicator. In some cases, this procedure has been known to result in pain and injury. Because of the invasive nature of the procedure, patients often refuse testing or withdraw during the collection process resulting in inadequate specimen procurement. In our effort to streamline the specimen collection process, our team has developed working prototypes of two specimen devices (a NP wash collection device and an Oral Capsule saliva collection device).

* The NP wash device is designed to irrigate the patient's nasopharyngeal passage with 3 ml of sterile saline and recollect the solution for testing. In our preliminary testing, the study device was successful in collecting RNase P from the nasal passages 100% of the time while achieving a mean Cycle Threshold (CT) value of 29.5. Participants in early studies also reported the study device to be more comfortable (0.3/10 pain) than the nasopharyngeal swab (8/10 pain).
* The Oral Capsule device is a soft-hollow device that is inserted into the mouth, overlying their molars. As the patient bites on the device, it generates an intermittent suction force which pulls saliva into the device's specimen chamber. In preliminary testing, the saliva collection device was successful in consistently collecting approximately 1 ml of saliva with 5-10 seconds of use.

The study design of this new protocol will allow the study investigators calculate the study devices' sensitivity and specificity for pathogen testing and test for antibody response from each respective specimen, along with improving enrollment rates. This study will enroll up to 1000 participants from a pool of ED patients who received a nasopharyngeal swab for PCR testing as part of their standard work up. Enrolled patients will provide four specimens 1) saliva drool specimen, 2) Oral Capsule saliva specimen, 3) NP wash specimen, and 4) finger stick serum specimen. Specimens 1, 2, 3 will undergo RPP PCR testing and COVID-19 antibody testing. Specimen 4 will undergo COVID-19 antibody testing. Patients can opt out of any of the four study specimen collection processes. Manufacturing of the NP Wash and the Oral Capsule devices is handled by the UNMC Department of Emergency Medicine fabrication lab. The NP wash study device is manufactured using fused deposition modeling (FDM) 3D printing technology with polylactic acid (PLA) printing material. The Oral Capsule device is manufactured using FDM 3D printing technology with polypropylene printing material. All study device will be sterilized via a cidex rinse, allowed to dry, then stored in a specimen bag. The NP wash device is designed to irrigate the user's nasopharyngeal cavity with 3 ml of sterile saline and recapture the irrigation solution into a specimen chamber as it drains back from their nose. The Oral Capsule device is designed to collect saliva via intermittent suction force generated within the device as the patient repeatedly bite on the device. With the implementation of our study devices we anticipate the following potential paradigm shifts in testing procedures: 1) minimizing the invasive nature of the procedure as a swab applicator is not utilized and 2) the procedure can be performed by a healthcare professional or solely by the patient, minimizing the risk of cross-infection to the healthcare professional. Nasopharyngeal irrigation is a common home remedy (neti-pots/bottles) for cold symptoms and is generally well tolerated by the user.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older presenting to the UNMC ED, or admitted from the UNMC ED with a non-research nasopharyngeal swab ordered.

Exclusion Criteria:

* None, if the inclusion criterion is met.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of respiratory pathogen infections in emergency department patients-nasophayngeal wash | 1 year
  Determine the incidence rate of respiratory pathogen infections in emergency department patients using a nasopharyngeal wash specimen by means of a polymerase chain reaction (PCR).
Incidence rate of respiratory pathogen infections in emergency department patients -saliva drool specimen | 1 year
  Determine the incidence rate of respiratory pathogen infections in emergency department patients using a saliva drool specimen by means of a polymerase chain reaction (PCR).
Incidence rate of respiratory pathogen infections in emergency department patients-oral capsule saliva specimen | 1 year
  Determine the incidence rate of respiratory pathogen infections in emergency department patients using an oral capsule saliva specimen by means of a polymerase chain reaction (PCR).

SECONDARY OUTCOMES:
Study survey and pain rating-nose swab procedure | 1 year
  Patient will be asked to complete a study survey and provide a pain rating of the nose swab procedure using a 0-10 pain scale (0 = no discomfort to 10 = a lot of discomfort).
Study survey and pain rating-nasopharyngeal wash procedure | 1 year
  Patient will be asked to complete a study survey and provide a pain rating of the nasopharyngeal wash procedure using a 0-10 (0 = no discomfort to 10 = a lot of discomfort).
Study survey and pain rating-oral capsule saliva collection procedure | 1 year
  Patient will be asked to complete a study survey and provide a pain rating of the oral capsule saliva collection procedure using a 0-10 pain scale (0 = no discomfort to 10 = a lot of discomfort).

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Nguyen, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Thanh Nguyen, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brendish NJ, Malachira AK, Armstrong L, Houghton R, Aitken S, Nyimbili E, Ewings S, Lillie PJ, Clark TW. Routine molecular point-of-care testing for respiratory viruses in adults presenting to hospital with acute respiratory illness (ResPOC): a pragmatic, open-label, randomised controlled trial. Lancet Respir Med. 2017 May;5(5):401-411. doi: 10.1016/S2213-2600(17)30120-0. Epub 2017 Apr 6. PMID 28392237
- [Background] Zumla A, Al-Tawfiq JA, Enne VI, Kidd M, Drosten C, Breuer J, Muller MA, Hui D, Maeurer M, Bates M, Mwaba P, Al-Hakeem R, Gray G, Gautret P, Al-Rabeeah AA, Memish ZA, Gant V. Rapid point of care diagnostic tests for viral and bacterial respiratory tract infections--needs, advances, and future prospects. Lancet Infect Dis. 2014 Nov;14(11):1123-1135. doi: 10.1016/S1473-3099(14)70827-8. Epub 2014 Sep 1. PMID 25189349
- [Background] Abad, X. Biocontainment in low income countries: a short discussion. Medical Safety & Global Health. 2018. 7(1), 1-3. DOI: 10.4172/2574-0407/1000139.
- [Background] Interim guidelines for collecting, handling, and testing clinical specimens from persons for coronavirus disease 2019 (COVID-19). Center for Disease Control and Prevention. 2020. Retrieved from: https://www.cdc.gov/coronavirus/2019-ncov/lab/guidelines-clinical-specimens.html.
- [Background] Daley P, Castriciano S, Chernesky M, Smieja M. Comparison of flocked and rayon swabs for collection of respiratory epithelial cells from uninfected volunteers and symptomatic patients. J Clin Microbiol. 2006 Jun;44(6):2265-7. doi: 10.1128/JCM.02055-05. PMID 16757636
- [Background] Fry DE. Pressure Irrigation of Surgical Incisions and Traumatic Wounds. Surg Infect (Larchmt). 2017 May/Jun;18(4):424-430. doi: 10.1089/sur.2016.252. Epub 2017 Mar 1. PMID 28437197
- [Background] Ball, S. Optimal pressures and irrigation techniques in small-animal wound management. Veterinary Nursing Journal. 2017. 32(11). 325-328.
- [Background] Barnes S, Spencer M, Graham D, Johnson HB. Surgical wound irrigation: a call for evidence-based standardization of practice. Am J Infect Control. 2014 May;42(5):525-9. doi: 10.1016/j.ajic.2014.01.012. PMID 24773788